CLINICAL TRIAL: NCT05892822
Title: Amyotrophic Lateral Sclerosis Registry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: yilong Wang (Other)
Responsible Party: Sponsor-Investigator, yilong Wang, Vice-President of Beijing Tiantan Hospital,Chief Scientist of Neurology Center, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Other Study IDs: KY2023-013-02
Record Dates: First submitted 2023-05-16; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — In order to explore unknown pathogenic genes and therapeutic targets, this study will collect patient genetics to construct a Chinese ALS gene spectrum and establish an iPSCs library.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amyotrophic Lateral Sclerosis: This study is an observational study without grouping.
  Interventions: Other: Amyotrophic Lateral Sclerosis

INTERVENTIONS:
Other: Amyotrophic Lateral Sclerosis — All ALS patients included in this group.

SUMMARY:
This study takes amyotrophic lateral sclerosis (ALS) patients as the main research object. Through collecting genetics, imaging and clinical symptoms for Exploratory research, we will construct the gene spectrum of ALS in China, explore unknown pathogenic genes, explore the characteristic image characteristics of ALS, and establish the iPSCs library of ALS, providing resources and basis for the research of pathogenesis and treatment targets of ALS.

DETAILED DESCRIPTION:
This study is a multicenter, prospective registration study that will follow up patients with clinically confirmed and suspected amyotrophic lateral sclerosis for a period of 2 years. A total of 1000 patients will be included to dynamically observe the changes in clinical symptoms and signs, imaging, electrophysiology, biomarkers, biological samples and so on, which will construct a genetic profile of ALS in China, explore the etiology and pathogenesis, and establish an iPSCs library, provide a basis for finding treatment targets.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤ 80 years old;
* Patients are diagnosed definite or probable ALS according to the Awaji diagnostic criteria;
* Sign an informed consent form.

Exclusion Criteria:

* Unable to cooperate with research or complete follow-up due to geographical or other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to include an estimated 1000 ALS patients in China.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Gene Mutation Characteristics of ALS in Chinese | day 1
  Constructing a Chinese ALS genetic information database by collecting genetic information from patients.
The disease development of ALS in the Chinese | month 24
  Record the progress of patients' clinical symptoms from baseline through 2-year follow-up.

SECONDARY OUTCOMES:
Exploring the imaging characteristics of ALS in the Chinese | day 1, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  Record the change of the patient's head MRI from baseline through follow-up every 3 months.
Establishing an iPSCs library for ALS in the Chinese | day 1
  100 fALS and clinically typical sALS were selected. Monocytes were isolated from peripheral blood collected at baseline, and Reprogramming into iPSCs to establish iPSCs library.
Analysis of the correlation between electrophysiology characteristics and imaging characteristics of ALS in Chinese | day 1, month 3, month 6, month 9, month 12, month 15, month 18, month 21, month 24
  Record the progression of the disease from an electrophysiological and imaging perspective by conducting electromyography and head MRI every 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiernan MC, Vucic S, Cheah BC, Turner MR, Eisen A, Hardiman O, Burrell JR, Zoing MC. Amyotrophic lateral sclerosis. Lancet. 2011 Mar 12;377(9769):942-55. doi: 10.1016/S0140-6736(10)61156-7. Epub 2011 Feb 4. PMID 21296405
- [Background] Meng L, Bian A, Jordan S, Wolff A, Shefner JM, Andrews J. Profile of medical care costs in patients with amyotrophic lateral sclerosis in the Medicare programme and under commercial insurance. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Feb;19(1-2):134-142. doi: 10.1080/21678421.2017.1363242. Epub 2017 Sep 11. PMID 28891333
- [Background] van Rheenen W, van der Spek RAA, Bakker MK, van Vugt JJFA, Hop PJ, Zwamborn RAJ, de Klein N, Westra HJ, Bakker OB, Deelen P, Shireby G, Hannon E, Moisse M, Baird D, Restuadi R, Dolzhenko E, Dekker AM, Gawor K, Westeneng HJ, Tazelaar GHP, van Eijk KR, Kooyman M, Byrne RP, Doherty M, Heverin M, Al Khleifat A, Iacoangeli A, Shatunov A, Ticozzi N, Cooper-Knock J, Smith BN, Gromicho M, Chandran S, Pal S, Morrison KE, Shaw PJ, Hardy J, Orrell RW, Sendtner M, Meyer T, Basak N, van der Kooi AJ, Ratti A, Fogh I, Gellera C, Lauria G, Corti S, Cereda C, Sproviero D, D'Alfonso S, Soraru G, Siciliano G, Filosto M, Padovani A, Chio A, Calvo A, Moglia C, Brunetti M, Canosa A, Grassano M, Beghi E, Pupillo E, Logroscino G, Nefussy B, Osmanovic A, Nordin A, Lerner Y, Zabari M, Gotkine M, Baloh RH, Bell S, Vourc'h P, Corcia P, Couratier P, Millecamps S, Meininger V, Salachas F, Mora Pardina JS, Assialioui A, Rojas-Garcia R, Dion PA, Ross JP, Ludolph AC, Weishaupt JH, Brenner D, Freischmidt A, Bensimon G, Brice A, Durr A, Payan CAM, Saker-Delye S, Wood NW, Topp S, Rademakers R, Tittmann L, Lieb W, Franke A, Ripke S, Braun A, Kraft J, Whiteman DC, Olsen CM, Uitterlinden AG, Hofman A, Rietschel M, Cichon S, Nothen MM, Amouyel P; SLALOM Consortium; PARALS Consortium; SLAGEN Consortium; SLAP Consortium; Traynor BJ, Singleton AB, Mitne Neto M, Cauchi RJ, Ophoff RA, Wiedau-Pazos M, Lomen-Hoerth C, van Deerlin VM, Grosskreutz J, Roediger A, Gaur N, Jork A, Barthel T, Theele E, Ilse B, Stubendorff B, Witte OW, Steinbach R, Hubner CA, Graff C, Brylev L, Fominykh V, Demeshonok V, Ataulina A, Rogelj B, Koritnik B, Zidar J, Ravnik-Glavac M, Glavac D, Stevic Z, Drory V, Povedano M, Blair IP, Kiernan MC, Benyamin B, Henderson RD, Furlong S, Mathers S, McCombe PA, Needham M, Ngo ST, Nicholson GA, Pamphlett R, Rowe DB, Steyn FJ, Williams KL, Mather KA, Sachdev PS, Henders AK, Wallace L, de Carvalho M, Pinto S, Petri S, Weber M, Rouleau GA, Silani V, Curtis CJ, Breen G, Glass JD, Brown RH Jr, Landers JE, Shaw CE, Andersen PM, Groen EJN, van Es MA, Pasterkamp RJ, Fan D, Garton FC, McRae AF, Davey Smith G, Gaunt TR, Eberle MA, Mill J, McLaughlin RL, Hardiman O, Kenna KP, Wray NR, Tsai E, Runz H, Franke L, Al-Chalabi A, Van Damme P, van den Berg LH, Veldink JH. Common and rare variant association analyses in amyotrophic lateral sclerosis identify 15 risk loci with distinct genetic architectures and neuron-specific biology. Nat Genet. 2021 Dec;53(12):1636-1648. doi: 10.1038/s41588-021-00973-1. Epub 2021 Dec 6. PMID 34873335
- [Background] Oskarsson B, Gendron TF, Staff NP. Amyotrophic Lateral Sclerosis: An Update for 2018. Mayo Clin Proc. 2018 Nov;93(11):1617-1628. doi: 10.1016/j.mayocp.2018.04.007. Epub 2018 Jul 4. PMID 30401437
- [Background] Sances S, Bruijn LI, Chandran S, Eggan K, Ho R, Klim JR, Livesey MR, Lowry E, Macklis JD, Rushton D, Sadegh C, Sareen D, Wichterle H, Zhang SC, Svendsen CN. Modeling ALS with motor neurons derived from human induced pluripotent stem cells. Nat Neurosci. 2016 Apr;19(4):542-53. doi: 10.1038/nn.4273. PMID 27021939
- [Background] Rowe RG, Daley GQ. Induced pluripotent stem cells in disease modelling and drug discovery. Nat Rev Genet. 2019 Jul;20(7):377-388. doi: 10.1038/s41576-019-0100-z. PMID 30737492